CLINICAL TRIAL: NCT00547261
Title: Phase I Dose Escalation and Pharmacokinetic Study of SSR97225 Administered as a 1 Hour IV Infusion D1 Every 3 Weeks (Arm A) or Administered as a 1hour IV Infusion D1, D8, D15 Every 3 Weeks (Arm B) in Patients With Refractory Solid Tumors
Brief Title: Phase I Dose Finding Study of SSR97225 Given in Patients With Refractory Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of supply of the investigational product.
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED5710
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Neoplasms
Keywords: solid tumor; antimitotic; tubulin binder
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Arm A (Experimental): 1 hour IV infusion D1
  Interventions: Drug: SSR97225
- Arm B (Experimental): 1 hour IV infusion D1, D8, D15
  Interventions: Drug: SSR97225

INTERVENTIONS:
Drug: SSR97225 — every 3 weeks

SUMMARY:
The purpose of this study is to determine the maximally tolerated dose and the dose limiting toxicity of this antimitotic, tubulin binding investigational drug for those patients who have failed standard anticancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic or locally advanced non-hematological cancer
* Patients with solid tumors refractory to therapy or for whom no therapy exists

Exclusion Criteria:

* Five or more prior chemotherapy lines for metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Patients having discontinued previous specific anti-cancer treatment
* Patients who have not recovered from all toxic effects from previous specific anti-cancer treatment (excluding alopecia)
* Patients with abnormal biological/hematological parameters, cardiac abnormalities or serious infection/intercurrent illness likely to jeopardize the patient's safety or the course of the protocol treatment
* No adequate birth control methods

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) and dose limiting toxicity (DLT) | Study period

SECONDARY OUTCOMES:
Pharmacokinetic profile, antitumor activity in patients with measurable disease, effect of drug on CYP3A4 activity | Study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States